CLINICAL TRIAL: NCT05804578
Title: Using a Liquid Biopsy to Monitor Metastatic Breast Cancer Treatment
Brief Title: Using a Blood Test to Monitor Metastatic Breast Cancer Treatment
Acronym: BEACON
Status: Recruiting | Type: Observational
Sponsor: Dr. Christopher Mueller (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Queen's University (Other)
Responsible Party: Sponsor-Investigator, Dr. Christopher Mueller, Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: 6037248; 486377 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Breast Cancer
Keywords: Liquid Biopsy; Treatment Response; Circulating Tumour DNA; DNA Methylation; Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected from participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to assess the effectiveness of the mDETECT breast cancer blood test at monitoring treatment response in women with metastatic breast cancer undergoing treatment.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in Canadian women. While survival rates for women with metastatic breast cancer have almost doubled in the last 20 years, the 5-year survival rate is about 25%. Currently, determining whether a breast cancer therapy is working is very difficult. Women undergo CT-scans every three months to assess the effectiveness of their therapy. If the chosen treatment is not effective, a patient would have been delayed in receiving a more effective treatment and will be exposed to the serious side effects of their ineffective treatment during this time.

The investigators have developed a blood test, called mDETECT, which is a DNA methylation-based liquid biopsy that targets multiple tumour specific hypermethylated regions on DNA. DNA shed from tumours travels through the blood stream and which can be collected through a blood draw and analyzed for breast cancer specific methylation patterns. The mDETECT breast cancer assay is sensitive and specific and has been proven to work well in detecting breast cancer in women with metastatic disease. This assay has been designed to work with all subtypes of breast cancer. Moreover, this blood test measures changes in the size of the tumour; therefore, it will work with any treatment.

The goal of this observational study is to assess the effectiveness of the mDETECT breast cancer blood test in women undergoing treatment for metastatic breast cancer to determine if a response to therapy can be seen earlier than the current 3 month time point for CT-scans. In this study, women undergoing treatment for metastatic breast cancer will be recruited. Participants will have blood drawn at baseline and multiple timepoints throughout treatment. The participants will also be monitored using the current standard of care, imaging every 3 months with CT-scans. The aim of this study will be to determine if the mDETECT blood test can predict within the first few weeks of treatment the results of the 3 month CT-scan.

ELIGIBILITY:
Inclusion Criteria

-Adult women (≥ 18 years of age) with proven diagnosis of adenocarcinoma of the breast with evidence of recurrent or metastatic disease not amenable to resection or radiation therapy with curative intent [to be herein described as 'metastatic']

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on both women with newly diagnosed metastatic breast cancer and women previously treated with metastatic breast cancer, regardless of treatment or breast cancer subtype.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in ctDNA level from baseline to 6 months of treatment | Baseline - 6 months
  The change in circulating tumour DNA methylation level over the course of treatment (Baseline blood draw, with timing of every standard of care blood draw for 8 weeks after treatment initiation, then monthly with standard of care blood draw for up to six after treatment initiation).
Changes in radiographic tumour assessments for monitoring response to treatment | 3 months and 6 months
  Radiographic tumor assessments will be performed as per RECIST v.1.1
Change in measurable lytic lesions in participants with bone only metastasis assessed by CT scans as measured per RECIST v.1.1 | 3 months and 6 months

SECONDARY OUTCOMES:
Progression-free survival in patients with increasing, stable, and decreasing ctDNA levels during treatment | Baseline - 6 months
  Progression-free survival is the time from enrolment in the study to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Mueller, Ph.D., Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Kingston Health Sciences Centre - Cancer Centre of Southeastern Ontario, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario